CLINICAL TRIAL: NCT03304847
Title: Arrhythmogenic Substrate Assessment in Patients With Primary Cardiomyopathies and/or Channellopaties With and Without History of Brugada Syndrome: A Prospective Follow-up Study
Brief Title: Arrhythmogenic Substrate in Primary Cardiomyopathies and/or Channellopathies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Chief of Arrhythmology Deartment, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSDonato 01-Cardiomyopathy
Record Dates: First submitted 2017-09-22; First posted 2017-10-09 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation (Other): Radio-frequency catheter ablation
  Interventions: Other: ablation

INTERVENTIONS:
Other: ablation — radio-frequency applications on arrhythmogenic substrate
  Other Names: radio-frequency ablation

SUMMARY:
This study assesses the value of arrhythmogenic substrate identification and elimination by catheter ablation to prevent recurrent ventricular arrhythmias and sudden cardiac death in a series of selected patients with primary cardiomyopathy and/or channellopaties with ICD implantation.

DETAILED DESCRIPTION:
The present study is designed as a prospective single center study. All selected patients with implanted ICD to prevent VT/VF recurrence who are referred to the Arrhythmology Department of San Donato Milanese Hospital, for the management of a primary cardiomyopathy fulfilling the inclusion criteria will be enrolled. Primary cardiomyopathies include: - dilated cardiomyopathy (DCM), - arrhythmogenic right ventricular cardiomyopathy (ARVC), - left ventricular non-compaction (LVNC), - early repolarization syndrome (ER), and - hypertrophic cardiomyopathy (HCM).Channellopaties incude - Long QT syndrome and J-wave syndrome) Patients with or without a family history of BrS, will also be included. Endo-epicardial electroanatomical 3Dmapping and RFA ablation will be systematically performed according to a standardized procedure. Patients will be monitored for at least 3 days after RF ablation. Before hospital discharge, echocardiography and 12-lead ECG will be performed. Patients will be followed-up clinically after the procedure as per normal clinical practice. Follow-up visits will be systematically scheduled at 3, 6, 12, 18 and 24 months. 12-lead ECG and ICD interrogation will be performed at each follow-up visit. Patients will be instructed to immediately contact the center in case of symptoms suggestive of ventricular arrhythmias. Documentation for intercurrent events will be requested and collected. The maximal duration of study participation for the individual patients is two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by cardiomyopathies and/or channellopaties (long QT syndrome and J-wave syndrome) with and without documented family history of BrS;
* Presence of symptoms attributable to VA and/or presenting documented arrhythmic episodes;
* Patients with an ICD already implanted;
* Patients referred to the centre for an electrophysiological study and indication for a potential concomitant radio-frequency catheter ablation (RFA) of ventricular tachycardia (VT) or ventricular fibrillation (VF);
* Age ≥ 18;
* Willingness to attend follow-up examinations;
* Written informed consent for the participation in the trial

Exclusion Criteria:

* Pregnancy or breast-feeding;
* Life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from ventricular fibrillation or ventricular tachycardia | two years
  Survival from recurrent ventricular arrhythmias

SECONDARY OUTCOMES:
Measurements of Areas of prolonged ventricular potentials obtained by electroamatomocal maps before and after ablation | 1 day
  Electrophysiological characterization of the arrhythmogenic substrate by electroanatomical maps

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — Chief of Arrhythmology Department
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No